CLINICAL TRIAL: NCT04838548
Title: An Open-Label, Multi-Cohort, Multi-center, Non-Randomized, Phase II Clinical Study to Evaluate the Efficacy and Safety of MRG003 in Patients With EGFR-Positive Advanced Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of MRG003 in Patients With EGFR-Positive Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG003-002
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: MRG003; Antibody Drug Conjugate (ADC); EGFR; Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG003 (Experimental): On the first day of every 3 weeks, MRG003 will be administered via intravenous infusion at 2.0 mg/kg calculated based on the actual body weight
  Interventions: Drug: MRG003

INTERVENTIONS:
Drug: MRG003 — Administered intravenously

SUMMARY:
The objective of this study is to assess the efficacy, safety of MRG003 as single agent in EGFR-positive advanced non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the ICF and follow the requirements specified in the protocol.
* Age: ≥18 years，both genders.
* Expected survival time≥6 months.
* Patients with histologically confirmed advanced non-small cell lung cancer, and without histologically confirmed small cell lung cancer (SCLC).
* Positive EGFR expression in tumor specimen.
* Failed in the prior second-line or above standard of care therapies.
* Archival or biopsy tumor specimens should be provided.
* Patients must have measurable lesions according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1).
* ECOG performance score 0 or 1.
* AEs related to prior systemic chemotherapy and radical/extensive radiotherapy have recovered to ≤ Grade 1 based on National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE V5.0).
* No severe cardiac dysfunction with left ventricular ejection fraction (LVEF) ≥ 50%.
* Organ functions and coagulation function must meet the basic requirements.
* Patients with childbearing potential must use effective contraception during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

* History of hypersensitivity to any component of the investigational product.
* No documented progression after prior treatment, or recurrence during or after prior treatment.
* Received radiotherapy, chemotherapy, biologicals, immunotherapy or other anti-tumor drugs within 4 weeks prior to the first dose of study treatment.
* Presence of central nervous system metastasis.
* Patients with significant clinical symptoms such as pleural, abdominal or pericardial effusion requiring puncture drainage prior to the first dose of study drug.
* Any severe or uncontrolled systemic disease judged by the investigator.
* Patients with poorly controlled heart diseases.
* Evidence of active infections, including Hepatitis B, Hepatitis C or human immunodeficiency virus (HIV) infection.
* Active bacterial, viral, fungal, rickettsial, or parasitic infection requiring systemic therapy.
* Prior history of other primary malignancies.
* History of the following ophthalmologic abnormalities: severve dry eye syndrome; keratoconjunctivitis sicca; severe exposure keratitis; any other condition that may increase the risk of corneal epithelial damage.
* History of severe skin disease requiring interruption of previous EGFR targeted therapy; or chronic skin disease requiring oral or intravenous therapy.
* History of interstitial lung disease (ILD) or pneumonitis, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.
* Pulmonary radiotherapy > 30 Gy within 6 months prior to first dose of study drug.
* Pulmonary embolism or deep vein thrombosis within 3 months prior to the first dose of study drug.
* Patients with active autoimmune disease or history of autoimmune disease, who are using immunosuppressive agents or systemic hormone therapy and still receiving within 2 weeks prior to enrollment.
* History of allogeneic tissue or solid organ transplant.
* Female patients with a positive serum pregnancy test or who are breast feeding or do not agree to take adequate contraceptive measures during the treatment and for 6 months after the last dose of study treatment.
* Active uncontrolled concomitant diseases that might limit patient's compliance with study requirements, or compromise patient's ability to provide written informed consent.
* Other conditions inappropriate for participation in this clinical trial, at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Investigator | Baseline to study completion, up to 12 months
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed by investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Baseline to study completion, up to 12 months
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Duration of Response (DoR) | Baseline to study completion, up to 12 months
  DOR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Time to Response (TTR) | Baseline to study completion, up to 12 months
  TTR is defined as the duration from the start of treatment to the first onset of CR or PR in tumor evaluation.
Disease Control Rate (DCR) | Baseline to study completion, up to 12 months
  DCR is defined as the proportions of patients achieving CR, PR, and stable disease (SD) after treatment.
Overall Survival (OS) | Baseline to study completion, up to 12 months
  OS is defined as the duration from the start of treatment to death of any cause.
Adverse Events (AEs) | Baseline to 60 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No